CLINICAL TRIAL: NCT06886984
Title: EFFECTS OF SOCIAL MEDIA REMINDERS ON ORAL HYGIENE MOTIVATION WITH FIXED ORTHODONTIC TREATMENT
Brief Title: Effects of Social Media on Oral Hygiene With Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Baris Baser, Associated Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KTU-DENT-BB-01
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Periodontal Inflammation; Orthodontic Appliance Complication
Keywords: oral hygiene; social media; fixed orthodontic treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social-media motivated group (Experimental): The patients assigned to social media group received two posts twice a week reminding hygiene procedures in addition to standardized oral hygiene instructions.
  Interventions: Behavioral: Social media motivation
- Non motivated group (No Intervention): The control group received only traditional communication including verbal and written instructions at the beginning of the therapy.

INTERVENTIONS:
Behavioral: Social media motivation — Reminding the oral hygiene instructions using social media tools to keep their oral hygiene stable
  Arms: Social-media motivated group

SUMMARY:
The aim of this study was to compare the efficacy of traditional and social media motivation strategies in improving oral hygiene with fixed orthodontic treatment.

DETAILED DESCRIPTION:
In this prospective, controlled clinical trial, 44 orthodontic patients were equally allocated to a social media (Facebook, Instagram and X (Twitter)) and control group. The control group received only traditional communication including verbal and written instructions at the beginning of the therapy. The patients assigned to social media group received two posts twice a week reminding hygiene procedures in addition to standardized oral hygiene instructions. Periodontal scores were obtained at 4-6-week intervals during six appointments (T1-T6) using the gingival index (GI), bleeding index (BI), and planimetric plaque quantification (PI) on photographs

ELIGIBILITY:
Inclusion Criteria:

* Class 1 malocclusion who had simple or moderate crowding and did not require tooth extraction.

Exclusion Criteria:

* Patients with functional appliances; surgical patients; those with a history of periodontitis, poor orthodontic hygiene, and/or physical or mental disabilities were excluded from the study.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Gingival Index | 6 months ( a score for every month)
  This is a clinical measurement. When the scores are higher, it means oral hygiene is getting worse.

SECONDARY OUTCOMES:
Bleeding Index | 6 months ( a score for every month)
  This is a clinical measurement. When the scores are higher, it means oral hygiene is getting worse.
Plaque Index | 6 months ( a score for every month)
  This is a combination of clinical and photographic measurement. When the scores are higher, it means oral hygiene is getting worse.

CONTACTS AND LOCATIONS:
Overall Officials: Barıs BASER, Assoc. Prof, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Faculty of Dentistry, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cimen E, Baser B. Effects of social media reminders on oral hygiene motivation with fixed orthodontic treatment: a randomized controlled trial. BMC Oral Health. 2025 Sep 29;25(1):1501. doi: 10.1186/s12903-025-06926-y. PMID 41023979